CLINICAL TRIAL: NCT04041167
Title: Impact of Lipoic Acid Use on Stroke Outcome After Reperfusion Therapy in Patients With Diabetes
Brief Title: Impact of Lipoic Acid Use on Stroke Outcome After Reperfusion Therapy in Patients With Diabetes (IMPORTANT)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Chosun University Hospital (Other); Chonbuk National University Hospital (Other); Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Kangho Choi, Study Director, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPORTANT
Record Dates: First submitted 2019-07-26; First posted 2019-08-01 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Stroke, Ischemic
Keywords: Reperfusion; Lipoic acid; Stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Thioctic Acid; Sodium Chloride; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alpha lipoic acid (Active Comparator): All patients will be assigned intravenous alpha lipoic acid 600mg within 24 hours of symptom onset. Patients will receive intravenous alpha lipoic acid 600mg/day for one week, followed by an oral pill of alpha lipoic acid 600mg/day for three months.
  Interventions: Drug: alpha lipoic acid
- Normal saline (Placebo Comparator): All patients will receive intravenous normal saline within 24 hours of symptom onset.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: alpha lipoic acid — alpha lipoic acid treatment
  Other Names: thioctacid
  Arms: Alpha lipoic acid
Drug: Saline — No alpha lipoic acid treatment
  Other Names: normal saline
  Arms: Normal saline

SUMMARY:
This study aims to investigate the effectiveness and safety of alpha-lipoic acid in patients with diabetes and ischemic stroke treated with reperfusion therapy.

DETAILED DESCRIPTION:
Despite significant advances in the prevention and treatment of stroke, it is still one of the leading causes of death and debilitating disease. Unfortunately, several neuroprotective strategies have failed in clinical trials. At present, it is reported that there are no pharmacological agents with putative neuroprotective actions that have demonstrated efficacy in improving outcomes after acute ischemic stroke (AIS) in humans. Previous stroke studies have confirmed that oxidative stress plays a vital role in stroke and in reperfusion following stroke. Therefore, the use of antioxidants could be a promising strategy for treating ischemia-reperfusion injury. Alpha-lipoic acid (aLA) is a potent antioxidant commonly used for the treatment of diabetic polyneuropathy (DPNP). The investigators previously demonstrated the neuroprotective and neurorestorative effects of aLA, mediated at least partially via insulin receptor activation, after cerebral ischemia in rats. Moreover, previous observational study of the investigators showed that patients with diabetes treated with aLA have better functional outcomes following AIS after reperfusion therapy than patients not using aLA.

Therefore, the investigators investigate whether patients with diabetes treated with aLA have better functional outcomes after AIS and reperfusion therapy than patients not treated with aLA in this prospective randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke within 6 hours of symptom onset
* Patients with diabetes
* Patients who underwent reperfusion therapy (Intravenous t-PA or endovascular thrombectomy)

Exclusion Criteria:

* Pre-existing disability (Modified Rankin Scale >= 1)
* Patients with severe renal disease (GFR <30 ml / min)
* Patients whose survival period is expected to be less than 12 months due to serious diseases such as terminal cancer or liver failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with functional independence | 3 months
  The modified Rankin Scale (mRS) consists of 7 levels, ranging from perfect health without symptoms (mRS score 0) to death (mRS score 6). We defined functional independence as mRS scores of 0-2 at 3 months after stroke.

SECONDARY OUTCOMES:
Rate of mortality | 3 months
  All cause of death within 3 months
Number of participants with BBB breakdown | 1 week
  Hemorrhagic transformation within 1 week, Brain edema at 1 week after stroke
Number of participants with early neurological deterioration | 2 weeks
  early neurological deterioration is defined as an increase of ≥1 point in motor power or an increase of ≥2 points in the total NIHSS score within 2 weeks
Number of participants with major bleeding | 3 months
  Intracranial and extracranial bleeding within 3 months
Number of participants with recurrence | 3 months
  Recurrent stroke within 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kangho Choi, MD, PhD, Principal Investigator — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hospital, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers.
Supporting Information: Study Protocol, CSR
Time Frame: We will share the data for one year after the end of the study.
Access Criteria: If a proposal for a joint research or a sub-study is proposed, the approval will be decided through a meeting of the committee.

REFERENCES:
- [Background] Choi KH, Park MS, Kim JT, Kim HS, Kim JH, Nam TS, Choi SM, Lee SH, Kim BC, Kim MK, Cho KH. Lipoic Acid Use and Functional Outcomes after Thrombolysis in Patients with Acute Ischemic Stroke and Diabetes. PLoS One. 2016 Sep 27;11(9):e0163484. doi: 10.1371/journal.pone.0163484. eCollection 2016. PMID 27677185
- [Background] Choi KH, Park MS, Kim HS, Kim KT, Kim HS, Kim JT, Kim BC, Kim MK, Park JT, Cho KH. Alpha-lipoic acid treatment is neurorestorative and promotes functional recovery after stroke in rats. Mol Brain. 2015 Feb 11;8:9. doi: 10.1186/s13041-015-0101-6. PMID 25761600